CLINICAL TRIAL: NCT02084134
Title: The Use of Perioperative Steroids in Patients Undergoing Transsphenoidal Resection of Pituitary Tumors or Cysts
Brief Title: Peri-Operative Steroid Management in Patients
Acronym: Steroid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201110174
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: Pituitary Adenoma; Pituitary Diseases
Keywords: pituitary adenoma; Pituitary Tumor; transsphenoidal resection; pituitary cyst
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases | interventions — Hydrocortisone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- steroid treatment arm (Active Comparator): Receives intravenous hydrocortisone 100mg and following surgery intravenous dexamethasone 0.5mg
  Interventions: Drug: hydrocortisone; Drug: dexamethasone
- non-steroid treatment (No Intervention): Subjects will not receive any steroids at the time of surgery or after surgery unless symptoms of adrenal insufficiency develop (i.e. nausea, vomiting, dizziness, or low blood pressure).

INTERVENTIONS:
Drug: hydrocortisone — 100mg at the time of surgery
  Other Names: intravenous hydrocortisone
  Arms: steroid treatment arm
Drug: dexamethasone — 0.5mg every 6 hours for a total of four doses
  Other Names: intravenous dexamethasone
  Arms: steroid treatment arm

SUMMARY:
During transsphenoidal resection of pituitary tumors and cysts, surgery is performed by a neurosurgeon and ear nose and throat surgeon. The pituitary tumor or cyst is reached by making a small hole in the back of the nose into the bottom of the skull. The surgeon is able to see the pituitary and tumor with an endoscope and remove the tumor through the hole.

Surgery on the pituitary can cause disruption in the secretion of ACTH and cause adrenal failure (lack of cortisol secretion) which can cause nausea, vomiting, low blood pressure, and rarely can be fatal. There is no consensus among endocrinologists and neurosurgeons about the use of perioperative steroids in pituitary patients. Traditionally, all patients undergoing pituitary surgery were given steroids before, during, and after surgery because of the assumption that there would be some compromise in the amount of ACTH released by the pituitary as a result of surgical trauma. Studies have failed to show, however, that ACTH secretion is in fact compromised during transsphenoidal pituitary microsurgery. As a result, there are some centers that routinely give perioperative steroids to all patients undergoing pituitary surgery and there are some centers that do not routinely give perioperative steroids. There are several retrospective and prospective studies that have addressed this issue and have shown that withholding perioperative steroids is safe, but there has never been a prospective study comparing the two approaches.

Objectives: The goal of this study is to prospectively compare two approaches to the perioperative management of patients undergoing transsphenoidal resection of a pituitary tumor or cyst. One protocol includes the routine use of perioperative steroids and the other does not. The investigators hypothesis, based on previous studies, is that patients who are adrenally sufficient do not routinely need to be treated with perioperative steroids. The investigators also hypothesize that the use of perioperative steroids may be associated with a higher rate of adverse outcomes

DETAILED DESCRIPTION:
Patients who are scheduled to undergo transsphenoidal resection for a pituitary tumor or cyst at the investigators institution will be screened prior to surgery for eligibility for this study. All patients deemed eligible will undergo a cosyntropin stimulation test to evaluate for adrenal insufficiency. Patients with adrenal insufficiency will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient with a pituitary adenoma or cyst (either non-functioning, prolactin secreting, growth hormone secreting, gonadotropin secreting, or TSH (Thyrotropin secreting hormone) scheduled to undergo transsphenoidal resection.

Exclusion Criteria:

* Patients with Cushing's Disease (pituitary tumor which secretes ACTH)
* Patients with a history of pituitary apoplexy (condition caused by hemorrhage into a pituitary adenoma which causes headache, double vision and hypopituitarism)
* Patients on long term glucocorticoid therapy
* Patients with adrenal insufficiency or who have not had their adrenal response evaluated prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-03; Primary Completion 2016-11-21 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M. Silverstein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Agha A, Liew A, Finucane F, Baker L, O'Kelly P, Tormey W, Thompson CJ. Conventional glucocorticoid replacement overtreats adult hypopituitary patients with partial ACTH deficiency. Clin Endocrinol (Oxf). 2004 Jun;60(6):688-93. doi: 10.1111/j.1365-2265.2004.02035.x. PMID 15163331
- [Background] Marko NF, Hamrahian AH, Weil RJ. Immediate postoperative cortisol levels accurately predict postoperative hypothalamic-pituitary-adrenal axis function after transsphenoidal surgery for pituitary tumors. Pituitary. 2010 Sep;13(3):249-55. doi: 10.1007/s11102-010-0227-6. PMID 20339931
- [Background] Marko NF, Gonugunta VA, Hamrahian AH, Usmani A, Mayberg MR, Weil RJ. Use of morning serum cortisol level after transsphenoidal resection of pituitary adenoma to predict the need for long-term glucocorticoid supplementation. J Neurosurg. 2009 Sep;111(3):540-4. doi: 10.3171/2008.12.JNS081265. PMID 19326985
- [Background] Hout WM, Arafah BM, Salazar R, Selman W. Evaluation of the hypothalamic-pituitary-adrenal axis immediately after pituitary adenomectomy: is perioperative steroid therapy necessary? J Clin Endocrinol Metab. 1988 Jun;66(6):1208-12. doi: 10.1210/jcem-66-6-1208. PMID 3372683
- [Background] Bhansali A, Dutta P, Bhat MH, Mukherjee KK, Rajput R, Bhadada S. Rational use of glucocorticoid during pituitary surgery--a pilot study. Indian J Med Res. 2008 Sep;128(3):294-9. PMID 19052341
- [Background] Inder WJ, Hunt PJ. Glucocorticoid replacement in pituitary surgery: guidelines for perioperative assessment and management. J Clin Endocrinol Metab. 2002 Jun;87(6):2745-50. doi: 10.1210/jcem.87.6.8547. PMID 12050244
- See also: Washington University School of Medicine, Research Participant Registry — https://vfh.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Steroid Treatment Arm | Non-steroid Treatment
Started | 23 | 20
Completed | 19 | 17
Not Completed | 4 | 3
Not completed — Protocol Violation | 4 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid Treatment Arm | Non-steroid Treatment | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 32
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 12 | 7 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adrenal Insufficiency
Description: Adrenal insufficiency was defined by a 30 or 60 min cortisol < 18 during a cosyntropin stimulation test
Time Frame: 6 weeks following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Treatment Arm | Non-steroid Treatment
Number analyzed (Participants) | 19 | 17
Participants | 2 | 1

2. Secondary Outcome: Percentage of Patients Discharged on Glucocorticoids
Description: Patient charts were reviewed to identify patients who were discharged on prednisone
Time Frame: 1 day (Day of hospital discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Treatment Arm | Non-steroid Treatment
Number analyzed (Participants) | 19 | 17
Participants | 8 | 2

ADVERSE EVENTS:
Arm/Group | Steroid Treatment Arm | Non-steroid Treatment
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid Treatment Arm (N=23) | Non-steroid Treatment (N=20)
Death (Immune system disorders) | 0 (0) | 1 (1) — One patient in non-steroid group died from meningitis which was not felt to be related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes